CLINICAL TRIAL: NCT01657422
Title: PACE+: Counseling Adolescents for Exercise and Nutrition
Acronym: PACEAdol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: San Diego State University (Other)
Responsible Party: Principal Investigator, Kevin Patrick, MD, MS, Kevin Patrick, MD, MS, Principal Investigaor and Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 7R01CA081495-04 (NIH)
Record Dates: First submitted 2012-07-27; First posted 2012-08-06 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Dietary Modification; Physical Activity
Keywords: Nutrition; Physical Activity; Adolescents
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PACE+ Intervention (Experimental): Intervention Group
  Interventions: Behavioral: PACE+
- Sun Protection (No Intervention): Control / Comparison group. Patients assigned to the comparison group will receive intervention strategies over a the course of 2 years including: (1) completion of a 30-minute office-based computer program resulting in on-screen feedback to address excess sun exposure prevention, and (2) 4 phone calls and 4 mailings over a 24-month period conducted by PACE+ staff members.

INTERVENTIONS:
Behavioral: PACE+ — Patients assigned to the intervention group will receive intervention strategies over a the course of 2 years including: (1) completion of a 45-minute office-based computer program resulting in an assessment and action plan for improvement in physical activity and nutrition behaviors; (2) a provider counseling session immediately following the computerized assessment, followed by (3) 12 phone calls and 24 mailings over a 24-month period conducted by PACE+ staff members
  Other Names: PACE+ Intervention
  Arms: PACE+ Intervention

SUMMARY:
PACE+ was developed to address the increased number of adolescents in our country that are at risk for cardiovascular disease, cancer, and other diseases due to inactivity, obesity, and malnourishment. PACE+ will evaluate the efficacy of an integrated clinical and home-based intervention to improve physical activity and nutrition behaviors in adolescents ages 11-15 over a period of 2 years.

This study is unique in that it will be one of the first to evaluate a combined physical activity and nutrition intervention for youth that revolves around the primary health care setting. The PACE+ intervention is particularly innovative in that three components - computer, provider counseling, and an extended home-based intervention - are unified through a common theoretical framework.

DETAILED DESCRIPTION:
Improved physical activity (PA) and nutrition behaviors in adolescents show great promise to reduce risk of cancers and other diseases. Fewer than 20% of adolescents meet recommendations for fat or fruits & vegetables consumption, and only 50% of adolescent girls and 67% of boys meet recommendations for vigorous PA. PACE+ will evaluate an integrated clinical and home-based intervention to improve physical activity (PA) and nutrition behaviors in adolescents. The intervention has three integrated components: a computer assessment and action planner; provider counseling; and 24 months of extended phone & mail contact. 768 male and female adolescents age 11 through 15; will be recruited from six healthcare settings. Subjects will be randomly assigned within practices to two successive one-year "doses" of PACE+ or a comparison condition involving counseling for sun protection behaviors. PACE+ assesses four behaviors: 1) dietary fat, 2) fruits & vegetable consumption, 3) physical activity, and 4) sedentary behavior. Primary behavioral outcomes, secondary outcomes, and selected mediators and process variables will be measured prior to the first office visit and at 6, 12 and 24 months. Primary outcomes will be measured by the 7-day physical activity recall and 3-day food record of fruits & vegetables and fat at 12 months. Secondary outcomes include adiposity, fitness, BMI, psychosocial mediators of change, and body image. Potential risks are psychological and physical, however the risks are slight and of low likelihood. Benefits include helping bring about healthier lifestyles to prevent weight gain and reduce premature morbidity and mortality due to cancer, cardiovascular disease and other health problems. This study will be the first to evaluate a combined physical activity and nutrition intervention for youth that revolves around the primary health care setting.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be in good general health and have the ability to read and speak English.

Exclusion Criteria:

* A known eating disorder,
* pregnancy,
* any cardiovascular or musculoskeletal problems that would limit their ability to comply with physical activity recommendations, and
* being in foster care (due to difficulty in obtaining follow-up measures).

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 819 (Actual)
Dates: Start 2000-08; Primary Completion 2004-11 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Dietary fat, fruits & vegetable consumption | 12months
  Equal in importance to the other two primary outcome measures, physical activity and sedentary behaviors
Physical activity | 12 months
  Equal in importance to the other two primary outcome measures, dietary fat, fruits and vegetables, and sedentary behaviors
sedentary behavior | 12 months
  equal in importance to the other two primary outcome measures: physical activity and diet fat, fruits and vegetable consumption

SECONDARY OUTCOMES:
dietary fat, fruits and vegetables | 24 months
  All were equal in terms of importance
physical activity | 24 months
sedentary behavior | 24 months

OTHER OUTCOMES:
weight status | 12 and 24 months
  Both time points equally important

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Patrick, MD, Principal Investigator — UCSD
Locations (2):
- United States (2):
  - University of California, San Diego, La Jolla, California
  - San Diego State University Foundation, San Diego, California